CLINICAL TRIAL: NCT06655532
Title: Effects of a Concurrent Training-based Exercise Program in Women Over 60 Years With Heart Failure With Preserved Ejection Fraction and Sarcopenia on Functional Capacity, Quality of Life and Cognitive Function
Brief Title: Effects of an Exercise Program in Women Over 60 yr. With HFpEF and Sarcopenia on Functional Capacity and Quality of Life
Acronym: TRAIN-SARC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRAIN-SARC
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure With Preserved Ejection Fraction (HFpEF); Sarcopenia; Women
Keywords: Heart Failure with Preserved Ejection Fraction; Sarcopenia; Cardiovascular Diseases; Heart Diseases; Heart Failure; Women
MeSH Terms: conditions — Sarcopenia; Cardiovascular Diseases; Heart Diseases; Heart Failure | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: This is a prospective study, blinded for the evaluator, 2 randomized groups (1:1) to receive standard management alone or combined with a program of training that will be carried out in a single centre.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Sham Comparator): Patients allocated to this arm will receive the standard medical treatment plus explicit recommendations for 12-week home-based moderate-intensity aerobic and strength training.
  Interventions: Behavioral: Usual Care
- Supervised aerobic plus moderate to high-intensity strenght training (Active Comparator): Patients allocated to this arm will receive the usual care plus supervised aerobic and moderate to high-intensity strength training.
  Interventions: Behavioral: Exercise Program

INTERVENTIONS:
Behavioral: Exercise Program — Patients allocated to this arm will receive the usual care plus supervised aerobic and moderate to high-intensity strength training twice weekly.
  Arms: Supervised aerobic plus moderate to high-intensity strenght training
Behavioral: Usual Care — Patients allocated to this arm will receive standard medical treatment plus explicit recommendations for 12-week home-based moderate-intensity aerobic and strength training. They will also receive a weekly phone call and an in-person monthly visit to monitor exercise training performance.
  Arms: Usual care

SUMMARY:
This prospective study will randomize (1:1) women with heart failure with preserved ejection fraction (HFpEF) and sarcopenia to receive standard management alone or a combined 12-week supervised exercise program (combining aerobic and strength exercise) carried out in a single centre.

After randomization, patients will be clinically evaluated. The primary endpoint (peakVO2) will be assessed by cardiopulmonary exercise testing (CPET) at 12 weeks. Women over 60 with HFpEF, functional class NYHA class II-III, and sarcopenia criteria will be enrolled. A sample size estimation [alfa: 0.05, power: 80%, a 20% loss rate, and at least a delta change of mean peakVO2: +1.9 mL/kg/min (SD±2)] of 40 patients (20 per arm) would be necessary to test our hypothesis.

DETAILED DESCRIPTION:
Heart failure with preserved ejection fraction (HFpEF) is a highly prevalent clinical entity that predominantly affects women, whose incidence has increased in the last decade and has a complex and multifactorial pathophysiology. Sarcopenia, a prevalent concurrent condition, appears to be associated with reduced muscle strength and reduced maximal functional capacity.

Supervised training programs in patients with heart failure with reduced ejection fraction and sarcopenia have improved functional capacity. However, the researchers do not have evidence about the effects of a supervised training program on patients with HFpEF and sarcopenia, mainly when affecting women older than 60. This work aims to evaluate the effect of a 12-week supervised exercise program in patients with HFpEF and sarcopenia on maximal functional capacity evaluated by peak oxygen consumption (peakVO2).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with heart failure with preserved ejection fraction according to 2021 ESC guidelines for Heart Failure, with N-terminal pro-B-type natriuretic peptide (NT-proBNP) >125 pg/mL, inthe last month.
* Stable symptomatic heart failure patients (New York Heart Association functional class II-III) during the last month.
* Age ≥ 60 years old.
* The participant is willing to give informed consent to participate in the study.
* SARC-F score ≥4 points.

Exclusion Criteria:

* Inability to perform a valid baseline cardiopulmonary exercise test.
* Cardiac pacemaker.
* Significant primary moderate-to-severe valve disease.
* Effort angina or signs of ischemia during CPET.
* Primary cardiomyopathies.
* Cardiac transplantation.
* Any other comorbidity with a life expectancy of less than one year.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-04 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Peak oxygen consumption | Primary outcome: Peak oxygen consumption will be evaluated at first visit and after 12 weeks. We will evaluate peak oxygen consumption change from baseline.
  Maximal functional capacity will be evaluated using incremental and symptom-limited cardiopulmonary exercise testing on a bicycle ergometer, beginning with a workload of 10 W and increasing gradually in a ramp protocol at 10-W increments every 1 minute. We define maximal functional capacity as when the patient stops pedalling because of symptoms and the respiratory exchange ratio (RER) was 1. During exercise, patients will be monitored with 12-lead electrocardiogram and blood pressure measurements every 2 minutes. Gas exchange data and cardiopulmonary variables were averages of values taken every 10 seconds. Peak oxygen consumption (PeakVO2) was defined as the highest value of VO2 during the last 20 seconds of exercise.

SECONDARY OUTCOMES:
Sarcopenia | Sarcopenia: SARC Questionnaire will be evaluated at first visit, after 12 weeks and after 16 weeks. We will evaluate the Sarc-F Questionnaire change from baseline.
  SARC-F (strength, assistance in walking, rise from a chair, climb stairs, and falls) it is a self-administered questionnaire that has five components: strength, assistance with walking, getting up from a chair, climbing stairs, and falls. It has a 3-level scoring system based on the level of difficulty, ranging from 0 (none) to 2 (very much), for each component.
Kansas City Cardiomyopathy Questionnaire Scales | The Kansas City Cardiomyopathy Questionnaire will be evaluated at first visit, after 12 weeks and after 16 weeks. We will evaluate the Kansas City Cardiomyopathy Questionnaire change from baseline.
  The Kansas City Cardiomyopathy Questionnaire includes 23 items that map to 7 domains: symptom frequency, symptom burden, symptom stability, physical limitations, social limitations, quality of life, and self-efficacy (the patient understanding of how to manage their heart failure). All Kansas City cardiomyopathy Questionnaire domains are scaled from 0 to 100, where scores represent health status as follows: 0 to 24, very poor to poor; 25 to 49, poor to fair; 50 to 74, fair to good; and 75 to 100, good to excellent. A change of 5 points is considered to be a small but clinically important change, whereas changes of 10 and 20 points are considered moderate-to-large and large-to-very-large clinical changes.

CONTACTS AND LOCATIONS:
Overall Officials: Laura López Bueno, PhD, Principal Investigator — Instituto de Investigacion Sanitaria INCLIVA
Locations (1):
- Hospital Clínico Universitario de Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No